CLINICAL TRIAL: NCT03586778
Title: Dry Needling for Patients With Back Pain: A Randomized Clinical Trial
Brief Title: Dry Needling for Patients With Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Concord Hospital (Other)
Collaborators: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Eric Gattie, Physical Therapist, Concord Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH lumbar needling
Record Dates: First submitted 2018-06-26; First posted 2018-07-16 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Back Pain
Keywords: Back Pain; Dry Needling
MeSH Terms: conditions — Back Pain | interventions — Dry Needling; Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment will be performed by an individual blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTEX-DN (Experimental): dry needling, manual therapy, and therapeutic exercise
  Interventions: Other: dry needling; Other: manual therapy; Other: therapeutic exercise
- MTEX (Active Comparator): manual therapy and therapeutic exercise
  Interventions: Other: manual therapy; Other: therapeutic exercise

INTERVENTIONS:
Other: dry needling — Dry Needling targeting the posterior musculature of the thoraco-lumbar spine and hips
  Arms: MTEX-DN
Other: manual therapy — Manual Therapy(mobilization/ manipulation) to address joint mobility of the thoraco-lumbar spine and hips
Other: therapeutic exercise — Exercise designed to improve performance of the paraspinal and abdominal musculature as well as the hip musculature. The exercise portion will also include a stretching program targeting the trunk and hip muscles which have been placed in a shortened position as a result of poor postures.

SUMMARY:
The aim of this trial will be to examine the short and long term effectiveness of dry needling on pain, disability, and patient perceived improvements in patients with back pain attending physical therapy. The investigators hypothesize that patients who receive dry needling, manual therapy, and exercise will achieve greater reductions in pain and disability in the short (6 weeks) and long term (6 and 24 months) compared to those who receive just manual therapy, and exercise.

DETAILED DESCRIPTION:
Background: Back pain is a very common and costly disorder. The financial burden is one of the highest of all health issues. Current treatments are not adequately effective for a large proportion of patients who continue to experience recurrent pain and ongoing disability. Therefore, new treatment strategies should be investigated in an attempt to reduce the disability and high costs associated with back pain.

Dry needling is a technique in which a fine needle is used to penetrate the skin, subcutaneous tissues, and muscle with the intent to mechanically disrupt tissue without the use of an anesthetic. Dry needling is emerging as a treatment modality that is widely used clinically to address a variety of musculoskeletal conditions. Recent studies of dry needling have shown decreased pain, increased pain pressure threshold, improved range of motion, and decreased disability in the short term. The majority of these studies examined dry needling using methods atypical to clinical practice (dry needling as a sole treatment, or fewer visits than is common practice). No studies have included long-term follow up. A clinical trial with realistic treatment time frames and methods consistent with clinical practice is needed to examine the effectiveness of dry needling on reducing pain and enhancing function in patients presenting with back pain. Both short and long term treatment outcomes need to be collected as there is emerging evidence that dry needling may be more effective in maintaining treatment effects in the long term. Therefore, the aim of this trial will be to examine the short and long term effectiveness of dry needling on pain, disability, and patient perceived improvements in patients with low back pain.

Purpose: The aim of this trial will be to examine the short and long term effectiveness of dry needling on pain, disability, and patient perceived improvements in patients with back pain.

Design: The investigators will conduct a randomized controlled trial in accordance with the CONSORT guidelines. All patients with back pain referred to physical therapy will be screened for eligibility criteria. Participants will be randomized to receive 1) dry needling, manual therapy, and exercise or 2) manual therapy and exercise. Participants will receive 8 treatments over a maximum of 6 weeks.

Methods: The primary outcome will be disability as measured by the Modified Oswestry Disability Index. Pain and patient perceived improvement will also be recorded. STarT Back clinical measurement tool will be used to monitor patient's risk dto develop chronic back pain. Outcome measures will be assessed at 6 weeks, 6 months, and 24-months by an assessor who is blind to the group allocation of the participants to determine the short and long-term treatment effects.

Data Analysis: The investigators will examine the primary aim with 2-way repeated-measures analysis of variance (ANOVA) with treatment group (MTEX vs. MTEX-DN) as the between subjects independent variables and time (baseline, 6 weeks, 6 months, 24 months) as the within-subjects independent variable. The hypothesis of interest is the 2-way group * time interaction.

Significance: The successful completion of this trial will provide evidence to demonstrate whether dry needling is effective for the management of back pain when used in a combined treatment approach as is commonly practiced clinically.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of back pain
* Modified Oswestry Disability Index > 10 points=20%

Exclusion Criteria:

* Red flags noted in the patient's Low Back Medical Screening (i.e. tumor, fracture, metabolic diseases, Rheumatoid Arthritis, prolonged history of steroid use, pregnancy, ankylosing spondylitis, cauda equina).
* Use of high doses of blood thinners
* Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the lower extremity, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
* Workers compensation or pending legal action regarding their back pain
* Insufficient English language skills to complete all questionnaires
* Inability to comply with treatment and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Modified Oswestry Disability Index(MODI) | baseline, six weeks, six months and 24 months
  Modified Oswestry Disability Index (MODI) is one of the modified versions of the Oswestry Disability Index. It consists of 10 items addressing different aspects of function. Each item is scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage.

SECONDARY OUTCOMES:
Change from baseline of Visual Analog Scale (VAS) | baseline, six weeks, six months and 24 months
  Visual Analog Scale (VAS) is a single item measure of pain using a 100 mm horizontal line anchored on the left side of which represents "no pain" and the right side represents "the worst pain imaginable". Patients mark a score by making a vertical line, where they feel it best represents their pain intensity.
Fear Avoidance Belief Questionnaire ( FABQ) | baseline, six weeks, six months and 24 months
  Fear Avoidance Belief Questionnaire ( FABQ) focused specifically on patients' beliefs about how physical activity and work affects their low back pain.
Global Rating of Change (GROC) | six weeks, six months and 24 months
  Global Rating of Change (GROC) is a 15-point scale used to quantify a patient's improvement with treatment or to record the clinical course of a condition over time. Patients are asked to describe their overall condition since the start of treatment until the present time with options ranging from -7 ("a very great deal worse") to +7 ("a very great deal better") and 0 being described as "about the same."
STarT Back | baseline, six weeks, six months and 24 months
  STarT Back is a clinical measurement tool is a questionnaire used to help to categorize patients into three subgroups based on their risk for developing chronic lower back pain. The STarT Back clinical measurement tool consists of 9 items including leg pain, common pain, disability (2 items), bothersomeness, catastrophization, fear, anxiety, and depression. Each question is answered on either a 5 point Likert scale or a 10 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian DG Sabadis, MS, Principal Investigator — Concord Hospital
Locations (1):
- Concord Hospital Rehabilitation Services, Concord, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No